CLINICAL TRIAL: NCT01329926
Title: Molecular Analysis of Adult Human-derived Neural Stem Cells
Brief Title: Molecular Analysis of Human Neural Stem Cells
Status: Withdrawn | Type: Observational
Why Stopped: insufficient funding
Sponsor: NeuroGeneration (Industry)
Responsible Party: Principal Investigator, Michel F. Levesque, MD, Principal Investigator, NeuroGeneration
Other Study IDs: NGN-9001
Record Dates: First submitted 2011-03-31; First posted 2011-04-06 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Parkinson's Disease; Parkinsonism
Keywords: Parkinson's disease; Neural stem cells
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tissue obtained during neurosurgical procedures yields undifferentiated neural stem cells that are subsequently expanded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neural stem cells
  Interventions: Procedure: Harvesting of neural stem cells

INTERVENTIONS:
Procedure: Harvesting of neural stem cells — During neurosurgical procedures, tissue samples are obtained along trajectory of implanted electrodes or removal of stimulators previously implanted.

SUMMARY:
The aim of this study is to develop and optimize methods to isolate, propagate and differentiate adult human neural stem cells from patients with degenerative neurological disorders like Parkinson's disease.

DETAILED DESCRIPTION:
In this project the investigators propose to analyze tissue samples from different nervous system regions obtained during neurosurgical procedures in order investigate the presence of neural stem cells in different cerebral areas. The investigators will also evaluate techniques for neural stem cell cryopreservation, for possible future therapeutic uses. Patients with degenerative neurological disorders like Parkinson's disease undergoing neurosurgical procedures meeting our selection criteria will be candidate for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent prior to study
2. Male or Female with Diagnostic Criteria of Parkinson's disease or neurodegenerative disorder undergoing a neurosurgical procedure
3. Age 35 to 85 years old
4. Parkinson's disease not due to trauma, infection, brain tumor, cerebrovascular disease
5. Hoehn and Yahr Stage III or IV
6. Parkinson's disease observed in the absence of:

   * Oculomotor palsy
   * Cerebellar sign
   * Orthostatic hypotension (drop greater than 20mmHg in mean pressure)
   * Pyramidal sign
   * Amyotrophy
7. Good general health or stable medical condition well controlled, without contraindications to anesthesia

Exclusion Criteria:

1. Patients with severe dementia and brain atrophy on MRI
2. Patients with severe hypertension; renal, liver, cardiac or other major organ disease; coagulopathy; cancer; other significant systemic illnesses; hepatitis, HIV
3. Patients older than 85 or younger than 35
4. Patients who withhold informed consent
5. Patients with a history of alcohol or drug abuse
6. Sexually active women of childbearing potential without adequate form of birth control
7. Evidence of abnormal coagulation or anticoagulant therapy
8. Pregnancy or lactation
9. History of seizure disorders or current use of antiepileptic medication
10. Severe cognitive impairment
11. Clinically significant laboratory abnormality

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease or parkinsonism
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06-30; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuronal differentiation into dopaminergic neurons | 6 months
  Differentiation of at least 10% of dopaminergic neurons is targeted as the primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Michel F Levesque, MD, Principal Investigator — Los Angeles Neurosurgical Institute
Locations (1):
- Los Angeles Neurosurgical Institute, Los Angeles, California, United States

REFERENCES:
- See also: Related Info — http://www.neurogeneration.com